CLINICAL TRIAL: NCT04050319
Title: ATI Evidence-based Guide Investigating Medical and Preventative Services: Sports Medicine, Athletic Training and Physical Therapy Treatment, Return to Sport, and Outcomes Registry
Brief Title: ATI Evidence-based Guide Investigating Medical and Preventative Services
Status: Enrolling by invitation | Type: Observational
Sponsor: ATI Holdings, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: SOR08012019
Record Dates: First submitted 2019-08-05; First posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Sport Medicine
Keywords: concussions; Fractures; Instability; Sprains; Strains
MeSH Terms: conditions — Fractures, Bone; Sprains and Strains | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Screening and diagnosis if injured — physical therapy
  Other Names: physical therapy

SUMMARY:
The investigators goal is to provide a mechanism that allows for a better understanding of athlete management from injury prevention through maintenance of health or development of injury and rehabilitation. The goal is to describe best practice for prevention and treatment to maximize return to health, sport, and patient reported outcomes following time. This includes collection of pre-existing risk factors, prevention program participation, treatment initiatives, functional outcomes measured by standardized and validated tools from the published literature. It incorporates comorbidities and patient demographic characteristics. All of these components come together to form a remarkably comprehensive picture of athlete health, influencing factors, and their associated outcomes.

DETAILED DESCRIPTION:
The investigators goal is to provide a mechanism that allows for a better understanding of athlete management from injury prevention through maintenance of health or development of injury and rehabilitation. The goal is to describe best practice for prevention and treatment to maximize return to health, sport, and patient reported outcomes following time. This includes collection of pre-existing risk factors, prevention program participation, treatment initiatives, functional outcomes measured by standardized and validated tools from the published literature. It incorporates comorbidities and patient demographic characteristics. All of these components come together to form a remarkably comprehensive picture of athlete health, influencing factors, and their associated outcomes.

Data are collected via the athletic training electronic medical record system EMR and integrated with data from the investigators proprietary EMR system and are genuine to the community through clinical process. The data are collected in real-time with athletes and patients and the scores are immediately provided to the providing athletic trainer and therapist as well as archived for later Registry and scientific use.

Subsequent reporting can be adjusted to any variable collected which yields robust insights as to athlete health. However, no PHI information will be available.

ELIGIBILITY:
Inclusion Criteria:

Active in an Organized Sports Team,

Exclusion Criteria: None

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Individuals receiving medical and/or preventative services when part of an organized sports team.
Sampling Method: Non-Probability Sample
Enrollment: 35000 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
DASH - Disabilities of the Arm, Shoulder, and Hand | through study completion, an average of 1 year
  Subjective

CONTACTS AND LOCATIONS:
Overall Officials: Chris Stout, PsyD, Study Chair — ATI
Locations (1):
- ATI, Bolingbrook, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
Aggregated non-Private Health Information and non-Health Insurance Portability and Accountability Act data would be made available upon request.